CLINICAL TRIAL: NCT02954965
Title: Enhancing Mood Among Graduate Students: Evaluation of a Brief, Phone-Administered Behavioral Intervention
Brief Title: Brief Mood Enhancement Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00074337
Record Dates: First submitted 2016-09-30; First posted 2016-11-04 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Stress, Psychological; Burnout, Professional
Keywords: graduate student; burnout; stress; mood
MeSH Terms: conditions — Stress, Psychological; Burnout, Professional; Burnout, Psychological

ARMS (3):
- Reward (Experimental): A brief, phone-administered intervention designed to help graduate students increase the number of pleasant and rewarding activities in their daily lives.
  Interventions: Behavioral: Reward
- Approach (Experimental): A brief, phone-administered intervention designed to help graduate students block procrastination and avoidance and to approach important activities they are currently avoiding.
  Interventions: Behavioral: Approach
- Monitoring (No Intervention): Participants will monitor their current behaviors, mood, and burnout with no directed intervention to change behavior

INTERVENTIONS:
Behavioral: Reward — Brief behavioral intervention (administered during a 45-minute phone call) that is designed to improve graduate student burnout by helping participants to identify activities that are rewarding and pleasurable and to integrate these activities into their schedule.
  Arms: Reward
Behavioral: Approach — Brief behavioral intervention (administered during a 45-minute phone call) that is designed to improve graduate student burnout by helping participants to identify activities that are challenging, but important to their long-term goals and values, and to integrate these activities into their schedule.
  Arms: Approach

SUMMARY:
The purpose of the current study is to test the efficacy of two brief, behavioral interventions intended to improve burnout among doctoral-level graduate students (n = 102). Specifically, individuals will be randomly assigned to one of three intervention conditions: 1) Reward: a brief intervention to help participants increase engagement in healthy and rewarding values-driven behaviors, 2) Approach: a brief intervention to help participants identify and decrease emotion-driven avoidance of important goals, or 3) Control: a control condition that involves monitoring only. Multilevel modeling will be used to assess changes in burnout, mood, and stress, following the interventions, controlling for participants' individual baseline levels of these variables.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in any in-person (not online) Ph.D. program in the state of North Carolina
* Demonstrating above average levels of burnout
* Has regular access to the Internet
* Has a Social Security Number
* Is able to read and understand English

Exclusion Criteria:

* Current mania or psychosis
* Current suicidal ideation
* Are currently in psychotherapy, have been in psychotherapy in the past 8 weeks, or are planning to start psychotherapy during the course of the 10-day study
* Have had any changes in psychiatric medications in the past 8 weeks, are not taking medications as prescribed or are planning to change medications during the course of the 10-day study
* Are currently taking benzodiazepines Pro Re Nata (PRN)
* Are under 18 years old

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2016-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in burnout, as measured by the School Burnout Inventory total score | baseline (day 0) and post-intervention (day 10)
  Self-report questionnaire assessing burnout
Change in stress, as measured by the Perceived Stress Scale total score | baseline (day 0) and post-intervention (day 10)
  Self-report questionnaire assessing stress

SECONDARY OUTCOMES:
Change in mastery, as measured by the Pearlin Personal Mastery Scale total score | baseline (day 0) and post-intervention (day 10)
  Self-report questionnaires assessing mastery
Change in avoidance, as measured by the Brief Experiential Avoidance Questionnaire total score | baseline (day 0) and post-intervention (day 10)
  Self-report questionnaires assessing avoidance
Change in mood, as measured by the Positive and Negative Affect Schedule total scores for Positive and Negative Affect | baseline (day 0) and post-intervention (day 10)
  Self-report questionnaire assessing mood
Change in reward, as measured by the Environmental Reward Observation Scale total score | baseline (day 0) and post-intervention (day 10)
  Self-report questionnaires assessing environmental reward
Change in behavioral activation, as measured by the Activation sub-scale of the Behavioral Activation for Depression Scale | baseline (day 0) and post-intervention (day 10)
  Self-report questionnaires assessing behavioral activation
Change in functional impairment, as measured by the Modified Work and Social Adjustment Scale total score | baseline (day 0) and post-intervention (day 10)
  Self-report questionnaire assessing functional impairment
Change in quality of life, as measured by the WHOQOL-BREF total score | baseline (day 0) and post-intervention (day 10)
  Self-report questionnaire assessing quality of life
Change in depression symptoms, as measured by the General Depression scale of the Inventory of Depression and Anxiety Symptoms | baseline (day 0) and post-intervention (day 10)
  Self-report questionnaire assessing depression symptoms
Change in mastery, as measured by the average of the daily Importance ratings of activities (0-10) on the Daily Activities Monitoring Form | baseline (days 0-3) and intervention (days 3-10)
  Self-report monitoring form describing activities during the day, how enjoyable they were, and how important they were
Change in avoidance, as measured by the total score of the Avoidance/Rumination sub-scale of the Behavioral Activation for Depression Scale | baseline (day 0) and post-intervention (day 10)
  Self-report questionnaire assessing avoidance and rumination
Change in environmental reward, as measured by the average of the daily Pleasure ratings of activities (0-10) on the Daily Activities Monitoring Form | baseline (days 0-3) and intervention (days 3-10)
  Self-report monitoring form describing activities during the day, how enjoyable they were, and how important they were

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States